CLINICAL TRIAL: NCT00756561
Title: Intratesticular Hormone Levels in Healthy Young Men
Brief Title: HOP-2A - Intratesticular Hormone Levels
Acronym: HOP-2A
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, John Amory, Professor, University of Washington
Other Study IDs: 34593-B
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Results first posted 2013-07-19 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-05

CONDITIONS: Healthy; Male Infertility; Prostate Disease
Keywords: Fine Needle Aspiration; Male Health; Male Contraception
MeSH Terms: conditions — Infertility, Male; Prostatic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum blood, testicular tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this investigational study is to find out what hormones are present in healthy male testicles using fine needle aspiration.

DETAILED DESCRIPTION:
We will collect a very small amount of fluid from each testicle. Participation will last up to 12 weeks. The study involves a minimum of 4 visits, the screening visit and procedure Day, fine needle aspiration of the testes (about 1-1.5 hours each) and two follow-up visits (about 30-45 minutes). Over the course of the study, you will have a little less than a 1/3-cup of blood drawn (roughly 2-3 tablespoons at each visit).

ELIGIBILITY:
Inclusion Criteria:

* males between 18 and 50 years of age
* sperm count greater than 20 million/ml, greater than 50% motility, and greater than 15% normal morphology
* in good general health based on normal screening evaluation (consisting of a medical history, physical exam, normal sperm count, normal serum chemistry, hematology and baseline T, LH, and FSH levels)
* body mass index ≥18 and ≤32 kg/m2
* must agree not to participate in another research study involving drug exposure for the duration of the study

Exclusion Criteria:

* men in poor general health, with abnormal blood results
* sperm counts <20 million/ml on two tests
* chronic, ongoing alcohol or drug abuse
* participation in a long-term male contraceptive study within the past three months
* history of testicular or scrotal surgery
* history of infertility
* abnormal testicular exam
* abnormal DRE
* chronic pain syndrome
* use of steroids, testosterone, or medications which might interfere with androgen metabolism including ketoconazole, glucocorticoids
* known bleeding disorder
* use of medications which may affect bleeding time (ongoing aspirin or anti-inflammatory use, coumadin)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy males
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John K Amory, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Page ST, Amory JK, Anawalt BD, Irwig MS, Brockenbrough AT, Matsumoto AM, Bremner WJ. Testosterone gel combined with depomedroxyprogesterone acetate is an effective male hormonal contraceptive regimen and is not enhanced by the addition of a GnRH antagonist. J Clin Endocrinol Metab. 2006 Nov;91(11):4374-80. doi: 10.1210/jc.2006-1411. Epub 2006 Aug 29. PMID 16940442
- [Background] Anawalt BD, Amory JK, Herbst KL, Coviello AD, Page ST, Bremner WJ, Matsumoto AM. Intramuscular testosterone enanthate plus very low dosage oral levonorgestrel suppresses spermatogenesis without causing weight gain in normal young men: a randomized clinical trial. J Androl. 2005 May-Jun;26(3):405-13. doi: 10.2164/jandrol.04135. PMID 15867009
- [Background] Coviello AD, Bremner WJ, Matsumoto AM, Herbst KL, Amory JK, Anawalt BD, Yan X, Brown TR, Wright WW, Zirkin BR, Jarow JP. Intratesticular testosterone concentrations comparable with serum levels are not sufficient to maintain normal sperm production in men receiving a hormonal contraceptive regimen. J Androl. 2004 Nov-Dec;25(6):931-8. doi: 10.1002/j.1939-4640.2004.tb03164.x. PMID 15477366
- [Background] Coviello AD, Matsumoto AM, Bremner WJ, Herbst KL, Amory JK, Anawalt BD, Sutton PR, Wright WW, Brown TR, Yan X, Zirkin BR, Jarow JP. Low-dose human chorionic gonadotropin maintains intratesticular testosterone in normal men with testosterone-induced gonadotropin suppression. J Clin Endocrinol Metab. 2005 May;90(5):2595-602. doi: 10.1210/jc.2004-0802. Epub 2005 Feb 15. PMID 15713727
- [Background] Page ST, Kalhorn TF, Bremner WJ, Anawalt BD, Matsumoto AM, Amory JK. Intratesticular androgens and spermatogenesis during severe gonadotropin suppression induced by male hormonal contraceptive treatment. J Androl. 2007 Sep-Oct;28(5):734-41. doi: 10.2164/jandrol.107.002790. Epub 2007 May 9. PMID 17494097
- [Background] Zhao M, Baker SD, Yan X, Zhao Y, Wright WW, Zirkin BR, Jarow JP. Simultaneous determination of steroid composition of human testicular fluid using liquid chromatography tandem mass spectrometry. Steroids. 2004 Oct-Nov;69(11-12):721-6. doi: 10.1016/j.steroids.2004.05.020. PMID 15579324
- [Background] Kalhorn TF, Page ST, Howald WN, Mostaghel EA, Nelson PS. Analysis of testosterone and dihydrotestosterone from biological fluids as the oxime derivatives using high-performance liquid chromatography/tandem mass spectrometry. Rapid Commun Mass Spectrom. 2007;21(19):3200-6. doi: 10.1002/rcm.3205. PMID 17764104
- [Result] Roth MY, Lin K, Amory JK, Matsumoto AM, Anawalt BD, Snyder CN, Kalhorn TF, Bremner WJ, Page ST. Serum LH correlates highly with intratesticular steroid levels in normal men. J Androl. 2010 Mar-Apr;31(2):138-45. doi: 10.2164/jandrol.109.008391. Epub 2009 Sep 24. PMID 19779211

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through news media (newspaper, website) and college campus bulletin boards in Seattle, WA, between September - December 2008. All visits were at the University of Washington, Seattle, WA.
Pre-assignment Details: 15 screened, 3 did not meet inclusion criteria (2 for abnormal semen parameters, 1 for abnormal liver function), 1 decided not to enroll, and 1 did not complete study procedures because of study end. Data analysis was performed on the first 10 of 11 subjects completing procedures.
Groups:
- Healthy Normal Males: Men, 18-50 years of age, in good health
Period: Overall Study
Arm/Group | Healthy Normal Males
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Normal Males
Number analyzed (Participants) | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  Between 18 and 50 years | 23 [21 to 32]
Sex/Gender, Customized [Number; unit: participants]
  Male | 10
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 25.9 [23.4 to 28.7]
Sperm concentration [Median (Inter-Quartile Range); unit: millions/mL] | 75 [28 to 133]
Luteinizing Hormone (LH) [Median (Inter-Quartile Range); unit: IU/L] | 3.7 [2.1 to 5.4]
Follicle Stimulating Hormone (FSH) [Median (Inter-Quartile Range); unit: IU/L] | 1.8 [1.4 to 2.5]
Serum Testosterone (T) [Median (Inter-Quartile Range); unit: ng/mL] | 3.0 [2.3 to 3.9]
Serum Dihydrotestosterone (DHT) [Median (Inter-Quartile Range); unit: ng/mL] | 0.20 [0.12 to 0.24]
Serum Estradiol (E2) [Median (Inter-Quartile Range); unit: ng/mL] | 0.025 [0.019 to 0.029]
Testis volume [Median (Inter-Quartile Range); unit: mL] — volume for left and right testis
  mL | 25 [20 to 25]

OUTCOME MEASURES:

1. Primary Outcome: Intratesticular Hormones in Normal Men
Description: Average between right and left testis for each subject and serum hormone concentration in 10 normal men
Time Frame: 6-weeks
Population: per protocol
Measure: Median (Inter-Quartile Range); unit: ng/mL
Groups:
- Intratesticular Concentration: Average intratesticular hormone concentration between right and left testis in 10 normal men
- Serum Concentration: Serum hormone concentration in 10 normal men
Arm/Group | Intratesticular Concentration | Serum Concentration
Number analyzed (Participants) | 10 | 10
ng/mL
  Testosterone | 486 [429 to 897] | 3.0 [2.3 to 3.9]
  Dihydrotestosterone | 3.7 [1.1 to 4.7] | 0.20 [0.12 to 0.24]
  Estradiol | 2.7 [1.3 to 3.4] | 0.025 [0.019 to 0.029]

ADVERSE EVENTS:
Time Frame: 4 months
Description: The first subject was screened 9/26/2008; the last subject exited 1/16/2009. Subjects in the study are asked about adverse events and concomitant medications at every visit.
Arm/Group | Healthy Normal Males
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 4/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Normal Males (N=11)
discomfort at lidocaine injection site (Reproductive system and breast disorders) | 1 (1) — reported discomfort from 11/5/08 to 12/2/08. Discomfort usually ends within a few days; this subject habitually bicycled 20 miles per day, and was advised to reduce bicycling for a short time.
bruised ribs (Musculoskeletal and connective tissue disorders) | 1 (1) — Subject is security officer and bruised ribs while restraining someone.
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Subjects did not take any medications for their colds.

LIMITATIONS AND CAVEATS:
Early termination of study leading to data analysis of the first ten of eleven men receiving aspirations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes